CLINICAL TRIAL: NCT01617486
Title: Achieving Energy Balance in Overweight Post Partum Teens
Brief Title: Achieving Energy Balance in Post Partum Teens
Acronym: BALANCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 201105325; 5R01CA121534 (NIH)
Record Dates: First submitted 2012-04-02; First posted 2012-06-12 (Estimated); Last update posted 2012-06-12 (Estimated); Status verified 2012-06

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BALANCE (Experimental)
  Interventions: Behavioral: BALANCE

INTERVENTIONS:
Behavioral: BALANCE — The intervention will focus on the replacement of 'obesogenic' patterns (such as high soda intake, excess portion size, and sedentary activity) with 'energy' patterns (such as water consumption, appropriate portion size, and walking).

SUMMARY:
This proposal will test Balance Adolescent Lifestyle Activities and Nutrition Choices for Energy (BALANCE), a multilevel intervention administered through Parents as Teachers (PAT) and designed to reduce overweight in postpartum teens. The intervention will focus on the replacement of 'obesogenic' patterns (such as high soda intake, excess portion size, and sedentary activity) with 'energy' patterns (such as water consumption, appropriate portion size, and walking).

ELIGIBILITY:
Inclusion Criteria:

* between 12 to 20 years of age
* less than 1 year post partum
* current participant in Parents as Teachers

Exclusion Criteria:

* currently pregnant

Ages: 12 Years to 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1325 (Actual)
Dates: Start 2007-01; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
BMI change at 6 month post assessment | Baseline and 6 month post assessment
  Postpartum adolescents in the intervention group who are at risk for overweight (85th-94th percentile BMI) or are overweight (equal to or greater than the 95th percentile) at baseline will have a change in BMI with a lower absolute BMI at 6 month post assessment than those in the control group
BMI change at 1 year post assessment | Baseline to 1 year post assessment
  Postpartum adolescents in the intervention group who are at risk for overweight (85th-94th percentile BMI) or are overweight (equal to or greater than the 95th percentile) at baseline will have a change in BMI with a lower absolute BMI at the 1 year post assessment than those in the control group

SECONDARY OUTCOMES:
reduce caloric intake | baseline and 6 month post test
  Our secondary hypotheses are that at the conclusion of the study (6 month post assessment) when compared to the control group, there will be a significantly greater proportion of postpartum adolescents in the intervention group who reduce caloric intake.
Engage in moderate intensity walking | Baseline and 6 month Post test
  Our secondary hypotheses are that at the conclusion of the study (6 month post assessment) when compared to the control group, there will be a significantly greater proportion of postpartum adolescents in the intervention group who increase moderate intensity walking.
Improve their knowledge of energy patterns | Baseline and 6 month Post test
  Our secondary hypotheses are that at the conclusion of the study (6 month post assessment) when compared to the control group, there will be a significantly greater proportion of postpartum adolescents in the intervention group who improve their knowledge of energy patterns.
Increase frequency of performance of energy patterns | Baseline and 6 month post test
  Our secondary hypotheses are that at the conclusion of the study (6 month post assessment) when compared to the control group, there will be a significantly greater proportion of postpartum adolescents in the intervention group who increase frequency of performance of energy patterns.

CONTACTS AND LOCATIONS:
Overall Officials: Debra Haire-Joshu, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States

REFERENCES:
- [Result] Haire-Joshu D, Yount BW, Budd EL, Schwarz C, Schermbeck R, Green S, Elliott M. The quality of school wellness policies and energy-balance behaviors of adolescent mothers. Prev Chronic Dis. 2011 Mar;8(2):A34. Epub 2011 Feb 15. PMID 21324248
- [Result] Haire-Joshu D, Schwarz C, Budd E, Yount BW, Lapka C. Postpartum teens' breakfast consumption is associated with snack and beverage intake and body mass index. J Am Diet Assoc. 2011 Jan;111(1):124-30. doi: 10.1016/j.jada.2010.10.009. PMID 21185974
- [Derived] Haire-Joshu DL, Schwarz CD, Peskoe SB, Budd EL, Brownson RC, Joshu CE. A group randomized controlled trial integrating obesity prevention and control for postpartum adolescents in a home visiting program. Int J Behav Nutr Phys Act. 2015 Jun 26;12:88. doi: 10.1186/s12966-015-0247-8. PMID 26112041